CLINICAL TRIAL: NCT04144985
Title: Eyelid Retraction Discomfort With Cotton Tipped Applicator, Unimanual and Speculum Intravitreal Injection Techniques: Eyelid Retraction Technique Randomized Comparison Trial (Eyelid RETRACT)
Brief Title: Comfort Comparison of Intravitreal Injection Eyelid Retraction Techniques
Acronym: Eyelid RETRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Joseph Raevis, Chief Ophthalmology Resident, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JJR223
Record Dates: First submitted 2019-10-17; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Intravitreal Injection; Pain
Keywords: Discomfort; Visual Analog Scale; Speculum; Eyelid retraction; Cotton tipped applicator; Eyelid Speculum; Unimanual eyelid retraction
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eyelid Speculum (Active Comparator): Eyelid retraction was performed with an eyelid speculum.
  Interventions: Other: Visual analog scale (VAS) of pain to evaluate the discomfort participants experience.
- Cotton Tipped Applicator (Experimental): Eyelid retraction was performed with the cotton tipped applicator eyelid retraction technique.
  Interventions: Other: Visual analog scale (VAS) of pain to evaluate the discomfort participants experience.
- Unimanual Eyelid Retraction (Experimental): Eyelid retraction was performed with the unimanual eyelid retraction method.
  Interventions: Other: Visual analog scale (VAS) of pain to evaluate the discomfort participants experience.

INTERVENTIONS:
Other: Visual analog scale (VAS) of pain to evaluate the discomfort participants experience. — Eyelid retraction was performed with one of the three methods (eyelid speculum, unimanual eyelid retraction or cotton tipped applicator assisted eyelid retraction) and participants were then asked to rate their discomfort during the procedure with a visual analog scale (VAS) of pain.

SUMMARY:
This study evaluated the discomfort associated with eyelid retraction during intravitreal injections. Participants had eyelid retraction with one of three methods: eyelid speculum, unimanual eyelid retraction method or with a cotton tipped applicator eyelid retraction technique. All participants were given a pain survey immediately after the injection to evaluate their discomfort level.

DETAILED DESCRIPTION:
Comfort is an important factor in compliance and satisfaction during medical care With the millions of intravitreal injections done each year, even small improvements in participants' experiences could lead to significant benefit. During the process eye injections, the method of eyelid retraction has been shown to be one of the most significant sources of discomfort.

Many ophthalmologists use an eyelid speculum to retract the eyelids, but potentially more comfortable methods exist. The purpose of our study was to test the comfort eyelid retraction with an eyelid speculum to that of the unimanual eyelid retraction method and a cotton tipped applicator eyelid retraction technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants receiving an intravitreal injection

Exclusion Criteria:

* iodine allergy
* prior ocular surgery other than uncomplicated cataract surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Pain Associated with Different Eyelid Retraction Technique | 1 minute
  Within one minute of the injection, the participant was given a standard 100mm long visual analog scale (VAS) and asked to rate their pain from 0mm (no pain) to 100mm (the worst pain) regarding the process of the intravitreal injection.

SECONDARY OUTCOMES:
Difference in Pain in Treatment Naive Participants | 1 minute
  Visual analog scale (VAS) of pain was compared between participant that had prior intravitreal injections and those that were treatment naive. Within one minute of the injection, the participant was given a standard 100mm long visual analog scale (VAS) and asked to rate their pain from 0mm (no pain) to 100mm (the worst pain) regarding the process of the intravitreal injection.
Associations of Hemoglobin A1c and Ocular Pain | 1 minute
  Visual analog scale (VAS) of pain was compared to participants with different hemoglobin A1c level. Within one minute of the injection, the participant was given a standard 100mm long visual analog scale (VAS) and asked to rate their pain from 0mm (no pain) to 100mm (the worst pain) regarding the process of the intravitreal injection.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Raevis, MD, Principal Investigator — Kings County Hospital Department of Emergency Medicine
Locations (1):
- Kings County Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No